CLINICAL TRIAL: NCT03471026
Title: Advanced MRI in Surgery for Posterior Fossa Tumours - Predicting Post-operative Paediatric Cerebellar Mutism Syndrome and Surgical Guidance to Avoid it
Brief Title: Advanced MRI for Posterior Fossa Tumours
Status: Completed | Type: Observational
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 17NI17
Record Dates: First submitted 2018-02-23; First posted 2018-03-20 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2020-12

CONDITIONS: Cerebellar Mutism; Posterior Fossa Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- pCMS+: Children undergoing infratentorial craniotomy for brain tumour resection whom develop pCMS will undergo pre-, post-operative and delayed follow-up advanced MRI sequences
  Interventions: Diagnostic Test: Advanced MRI sequences
- pCMS-: Children undergoing infratentorial craniotomy for brain tumour resection whom do not develop pCMS will undergo pre-, post-operative and delayed follow-up advanced MRI sequences
  Interventions: Diagnostic Test: Advanced MRI sequences
- Controls: Healthy control children whom have never undergone intracranial surgery have had advanced MRI sequences acquired
  Interventions: Diagnostic Test: Advanced MRI sequences

INTERVENTIONS:
Diagnostic Test: Advanced MRI sequences — Structural, diffusion and perfusion MRI sequences

SUMMARY:
Post-operative paediatric cerebellar mutism syndrome (pCMS) is a well-recognised complication of resective surgery for brain tumours of the cerebellum and fourth ventricle in children. Occurring in around 25% of infratentorial craniotomies, it is characterised by a delayed onset of mutism and emotional lability, and may comprise motoric and cognitive cerebellar deficits. Transient mutism gives way to prolonged, and often incomplete, recovery. Neuroimaging studies are beginning to reveal anatomical and functional aberrancies in the brain of children with pCMS. The cerebellar efferent pathways are likely to be implicated as a neuroanatomical substrate in the development of pCMS, as shown by a handful of diffusion tractography studies to date. However, the pathophysiology of this condition still remains unclear. Hypoperfusion of supratentorial cortical and subcortical structures may mediate the speech and behavioural deficits seen in pCMS, and is a candidate for a causal pathophysiological mechanism.

This study aims to prospectively image children with pCMS using advanced MRI techniques including diffusion tractography and arterial spin labelling, and to correlate this with clinical descriptions of the syndrome.

All children referred to Great Ormond Street Hospital for Children with a posterior fossa brain tumour will be imaged pre-operatively, post-operatively and at delayed follow-up. In tandem with this, clinical assessments will be made of children post-operatively to ascertain which patients develop pCMS. In addition, anonymised advanced MRI data on healthy controls will be used as a comparator group.

ELIGIBILITY:
Inclusion Criteria:

Age <18 Referred and operated upon within study period Brain tumour of cerebellum, IVth ventricle, brainstem undergoing craniotomy for resection (including re-do surgery) No restrictions as to tumour histology or grade (embryonal tumour / glioma / ependymoma) Informed consent given by parents

Exclusion Criteria:

Non-neoplastic infratentorial lesions Claustrophobia Contraindication to MRI Pregnant female Scans missing at >2 timepoints Tumour resection surgery at another hospital if no pre- or post-operative scans available

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All children referred to our institution with a brain tumour of the posterior fossa
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2021-04-07 (Actual)

PRIMARY OUTCOMES:
Diffusion MRI tractography | 1 year
  To compare diffusion MRI derived tractography of the fronto-cerebellar circuitry (and associated metrics of fractional anisotropy and mean diffusivity) between patients with and without pCMS.
Arterial Spin Labeling Perfusion MRI | 1 year
  To compare cerebral blood flow (a metric derived from perfusion MRI) in frontal lobe regions between patients with and without pCMS.

SECONDARY OUTCOMES:
Clinical measure of severity of pCMS | 1 year
  CMS Severity Score (Robertson 2006 JNS Peds 105: 444-451):
  Clinical diagnosis of pCMS Yes / No
  If yes:
  Time of onset
  1. immediately post op
  2. Days 1-2
  3. Days 2-4
  4. => Day 4
  Mutism
  1. Mild (<1wk)
  2. Moderate (1-4wks)
  3. Severe (>4wks)
  Ataxia
  1. Mild (<1wk)
  2. Moderate (1-4wks)
  3. Severe (>4wks)
  Hypotonia
  1. Mild (can sit or stand by <1wk)
  2. Moderate (can sit or stand by 1-4wks)
  3. Severe (can sit or stand by >4wks)
  Irritability
  1. Mild (<1wk)
  2. Moderate (1-4wks)
  3. Severe (>4wks)
  Severe = at least 2 severe features Moderate = at least 2 moderate features or 1 moderate and 1 severe Mild = anything less than above

CONTACTS AND LOCATIONS:
Overall Officials: Chris Clark, PhD, Principal Investigator — University College London Institute of Child Health; Kristian Aquilina, MD, FRCS, Principal Investigator — Great Ormond Street Hospital; Sebastian M Toescu, MBChB (Hons), Principal Investigator — University College London Institute of Child Health
Locations (1):
- Great Ormond Street Hospital for Children, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Toescu SM, Hales PW, Cooper J, Dyson EW, Mankad K, Clayden JD, Aquilina K, Clark CA. Arterial Spin-Labeling Perfusion Metrics in Pediatric Posterior Fossa Tumor Surgery. AJNR Am J Neuroradiol. 2022 Oct;43(10):1508-1515. doi: 10.3174/ajnr.A7637. Epub 2022 Sep 22. PMID 36137658